CLINICAL TRIAL: NCT02285413
Title: Immunochemotherapy: Do Platin-based Chemotherapeutics Enhance Dendritic Cell Vaccine Efficacy in Melanoma Patients?
Brief Title: Platin-based Chemotherapeutics to Enhance Dendritic Cell Vaccine Efficacy in Melanoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL32381.000.10
Record Dates: First submitted 2013-05-11; First posted 2014-11-07 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Melanoma
Keywords: Melanoma; Dendritic cells; Cisplatin; Vaccine; Immunotherapy
MeSH Terms: conditions — Melanoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DC vaccination (Experimental): mature DC injected intradermally and intravenously loaded with mRNA encoding tumor-associated antigens gp100 and tyrosinase
  Interventions: Biological: DC vaccination
- DC vaccination with cisplatinum (Experimental): mature DC injected intradermally and intravenously loaded with mRNA encoding tumor-associated antigens gp100 and tyrosinase. each DC vaccine will be preceded by cisplatin infusion: 50 mg/m2, 1-2h before DC injection.
  Interventions: Biological: DC vaccination with cisplatinum

INTERVENTIONS:
Biological: DC vaccination — DC vaccination without cisplatinum
  Arms: DC vaccination
Biological: DC vaccination with cisplatinum — DC vaccination with cisplatinum
  Arms: DC vaccination with cisplatinum

SUMMARY:
This is an exploratory study and the primary objective is the immunogenicity and feasibility of combined chemotherapy-DC vaccination. The secondary objectives are the toxicity and clinical efficacy. This study will provide important data on the immunological efficacy of DC immunochemotherapy.

DETAILED DESCRIPTION:
1. Rationale Investigators have explored immunotherapy and have now vaccinated well over 200 stage III and IV melanoma patients in the Netherlands with monocyte-derived dendritic cell (DC) vaccines and proved that DC therapy is safe with minimal side effects.

   Cytotoxic chemotherapy and radiotherapy have long been viewed as strategies that directly impact the viability of the tumor cell, and that the immune system contributed little to their efficacy. The commonly held opinion was that chemotherapy and immunotherapy could not be combined because of the myelo-suppressive effect of most chemotherapeutic agents. However, it becomes increasingly obvious that chemotherapy also possess the capacity to trigger tumor antigen release and danger signals in a manner that provokes engagement of innate and adaptive immunity that may be capitalized upon.

   Small proof-of-concept clinical trials in cancer patients indicate that the efficacy of anti-cancer vaccines may indeed be enhanced by chemotherapy [2]. Also preliminary observations indicate that chemotherapeutic agents, in particular platinum compounds (cisplatin, carboplatin and oxaliplatin) are immunogenic and may contribute to reverse tumor cell induced immunosuppression/immune deviation.

   Investigators hypothesize that DC vaccination, when combined with other more conventional anti-tumor treatments such as chemotherapy, that eradicate large numbers of cancer cells, may allow the T cells to clear the remaining cancer cells and to provide immunological memory to prevent relapse.
2. Objectives This is an exploratory study and the primary objective is the immunogenicity and feasibility of combined chemotherapy-DC vaccination. The secondary objectives are the toxicity and clinical efficacy. This study will provide important data on the immunological efficacy of DC immunochemotherapy.
3. Study design This study is an open label randomized phase II study.
4. Study population Our study population consists of melanoma patients, with expression of melanoma associated tumor antigens gp100 and tyrosinase. Melanoma patients with regional lymph node metastasis in whom a radical lymph node dissection is performed within 2 months of inclusion in this study (further referred to as stage III) and melanoma patients with measurable distant metastases (further referred to as stage IV) will be included.
5. Main study endpoints The primary objective of the study is to investigate the immunogenicity and feasibility of combined chemotherapy-DC vaccination. The secondary objective is to investigate the toxicity and clinical responses (only in stage IV) upon DC immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

All patients:

* histologically documented evidence of melanoma
* stage III or IV melanoma according to the 2001 AJCC criteria
* melanoma expressing gp100. Tyrosinase is not mandatory but will be assessed.
* WHO performance status 0-1 (Karnofsky 100-70)
* life expectancy ≥3 months
* age 18-70 years
* no clinical signs or symptoms of CNS metastases
* WBC >3x10^9/l, lymphocytes >0.8x10^9/l, platelets >100x10^9/l, serum creatinine <150 µmol/l, serum bilirubin <25 µmol/l
* normal serum LDH (<450 U/l)
* expected adequacy of follow-up
* no pregnant or lactating women
* written informed consent

and in addition: Stage III melanoma

* radical regional lymphnode dissection is performed Stage IV melanoma
* at least one unidimensional measurable target lesions according to RECIST, not previously irradiated, and no significant symptoms of disease requiring other palliative treatments

Exclusion Criteria:

* any prior chemotherapy, immunotherapy or radiotherapy is allowed if completed more than 4 weeks prior to planned vaccination
* history of any second malignancy in the previous 5 years, with the exception of adequately treated basal cell carcinoma or carcinoma in situ of the cervix
* serious active infections, known HbsAg or HIV positive, or autoimmune diseases or organ allografts
* concomitant use of immunosuppressive drugs
* known allergy to shell fish (since it contains KLH)
* rapidly progressive symptomatic disease
* any serious clinical condition that may interfere with the safe administration of DC

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-02; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: number of participants with KLH and/or tumor-specific antigens immune responses. | 5 years
Feasibility: % of vaccines meeting the release criteria. | 5 years

SECONDARY OUTCOMES:
Toxicity: number of Participants with Adverse Events. | 5 years
Progression-free survival | 5 years
Overall survival | 5 years
Best objective response (only in stage IV) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Winette van der Graaf, professor, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands